CLINICAL TRIAL: NCT06484374
Title: A Study of Minimally Invasive Surgical Strategies for Robot-assisted Supratentorial Large Hematoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Affiliated Hospital of Nantong University (Other); The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SQ2023AAA030147
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Hematoma Brain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Craniotomy (Sham Comparator): Traditional craniotomy, by opening the skull and thus removing the hematoma
  Interventions: Procedure: Robot-assisted minimally invasive treatment
- Robot-assisted minimally invasive treatment (Experimental): Minimally invasive hematoma removal with robotic assistance
  Interventions: Procedure: Robot-assisted minimally invasive treatment

INTERVENTIONS:
Procedure: Robot-assisted minimally invasive treatment — An automatic surgical path planning system using artificial intelligence fused with neuroimaging is used to determine the surgical incision and drilling points; the principles followed include but are not limited to: avoidance of important functional areas such as language and motor cortex; avoidance of vascular densely populated areas; and individualized optimal paths for the three-dimensional morphology of the hematoma and spatial orientation.

SUMMARY:
The AI robot is used to design precise coordinates and access routes for hypertensive cerebral hemorrhage patients with large supratentorial hematomas in conjunction with imaging data, to clarify the therapeutic efficacy of robotic-assisted endoscopic debridement of precise minimally invasive surgical system for perioperative and long-term functional recovery of supratentorial hematomas, and to ultimately achieve the improvement of prognosis for this group of patients, and to alleviate the economic burdens on the society and the families

DETAILED DESCRIPTION:
In this randomized controlled study, we investigated the efficacy of robotic assistance for supratentorial large hematomas by comparing robotic-assisted minimally invasive removal of supratentorial large hematomas with conventional surgical hematoma removal. Our main comparisons were the 6-month mortality rate and good prognosis rate, and the main evaluation indexes included mRS score and GOS score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed by imaging (CT, CTA, etc.), measured by the ABC/2 method, and clearly recognized as having a supratentorial hypertensive cerebral hemorrhage.

   Patients with hematoma volume >30mL and GCS score ≥5;
2. The patient's age is 18-70 years old; Patients aged 18-70 years;
3. Time from onset to surgery ≤72h;
4. Repeat CT scan at least 6 hours after the diagnostic CT scan showed that the hematoma was stable;
5. SBP <180 mmHg was recorded near the time of random assignment;
6. mRS score ≤1 in the past medical history;
7. Patient/family informed and signed informed consent.

Exclusion Criteria:

1. The hematoma is not located on the curtain or the volume of the hematoma is less than 30 ml;
2. The onset of the disease is more than 3 days at the time of admission; Secondary cerebral hemorrhage (secondary causes such as aneurysm, vascular malformation, hemorrhagic transformation of cerebral infarction, tumor, trauma, drug-related or abnormal coagulation mechanism).
3. secondary causes such as aneurysm, vascular malformation, hemorrhagic transformation of cerebral infarction, tumor, trauma, drug-related or abnormal coagulation mechanism);
4. Presence of serious immune diseases (e.g., cirrhosis, malignant tumors, rheumatic immune diseases, etc.);
5. Poor compliance or inappropriate for enrollment as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Good prognosis rate after 6 months of follow-up | 6 months
  Good prognosis rate after 6 months of follow-up

IPD SHARING:
Plan to Share IPD: No